CLINICAL TRIAL: NCT01549431
Title: A Phase I Study of the Combination of Panobinostat and Carfilzomib in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study of the Combination of Panobinostat & Carfilzomib in Patients With Relapsed &/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Multiple Myeloma Research Consortium (Network); Novartis (Industry); Onyx Therapeutics, Inc. (Industry); Amgen (Industry); University of California, San Francisco (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Jonathan Kaufman, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00049368; WCI2011-11/MMRC036 (Other: Other)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat; carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combo of Panobinostat and Carfilzomib (Experimental): A cycle of therapy is 4 weeks (28 days in duration). Carfilzomib (with dexamethasone during cycle 1) will be administered intravenously infusion on days 1, 2 and 8, 9 and 15, 16 of every 28 day cycle. Panobinostat is administered orally three times per week.
  Interventions: Drug: Panobinostat; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Panobinostat — Panobinostat will be supplied as 5-mg or 20-mg pink/opaque-colored, hard gelatin capsules. Panobinostat is administered orally three times per week.
  * Standard 3+3 design
  * 3 out of 4 weeks
  Other Names: LBH589
Drug: Carfilzomib — Carfilzomib in Cycle 1 will be initiated intravenously at 20 mg/m² on Days 1 and 2 and escalated to 27 mg/m² for Days 8, 9, 15, and 16 of Cycle 1 and for the duration of treatment.
  * Standard 3+3 design
  * Days 1/2, 8/9 and 15/16 every 4 weeks
  Other Names: Kyprolis
Drug: Dexamethasone — Dexamethasone (4 mg) must be given prior to each carfilzomib infusion during Cycle 1. Dexamethasone pre-dose should continue through Cycle 2 if fever is observed post-dose, Cycle 2 Day 1, or thereafter associated with the infusion of carfilzomib.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of panobinostat and carfilzomib have on the patient's cancer. It will determine the side effects of different dose levels of panobinostat and carfilzomib and determine the best dose and schedule of the two drugs to recommend for future studies. The study will assess the effects of the drug on multiple myeloma. In addition, tests to study the way the drugs work will also be done.

The combination of the 2 drug classes have shown both pre-clinical (studies done in the lab) and clinical (studies done with people) effects against multiple myeloma. For this reason, these 2 drugs are being studied in combination to determine the side effects and anti-myeloma effects of the 2 drugs.

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase I study of panobinostat, carfilzomib in patients with relapsed/refractory multiple myeloma. Based on the preclinical data supporting the use of combined histone de-acetylase (HDAC) and proteasome inhibition, the incidence of single-agent panobinostat and carfilzomib anti-myeloma activity, and clinical data demonstrating safety and efficacy of panobinostat with a different proteasome inhibitor (bortezomib), this study will evaluate the combination of panobinostat and carfilzomib in patients with relapsed/refractory multiple myeloma in a phase I trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old
2. Diagnosis of multiple myeloma (MM) following at least one prior therapy; there is no maximum number or prior therapies
3. Patients must have relapsed/ refractory disease and be in need of therapy with evidence of measurable disease defined as at least one of the following:

   * Serum M protein ≥ 0.5 g/dl (≥ 5g/l)
   * Urine M protein ≥ 200 mg/24 hours
   * Serum free light chain (FLC) assay: Involved FLC assay ≥ 10 mg/dl (≥100 mg/l) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
   * Measurable plasmacytoma (Prior biopsy is acceptable)
4. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
5. Patients must meet the following laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 10⁹/L (growth factors cannot be used within 3 days of screening)
   * Hemoglobin ≥ 8 g/dl (PRBC transfusions cannot be used within 3 days of screening)
   * Platelets ≥ 75 x 10⁹/L (platelet transfusions cannot be used within 3 days of screening)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum potassium ≥ lower limit of normal (LLN)
   * Total serum calcium [corrected for serum albumin] or ionized calcium ≥ LLN. (treatment of hypercalcemia is allowed and subjects may enroll if hypercalcemia returns to normal with standard treatment)
   * Serum magnesium ≥ LLN
   * Serum phosphorus ≥ LLN
   * Creatinine clearance ≥ 30 ml/min (Cockcroft-Gault calculation)
   * Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
6. Baseline multigated acquisition scan (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
8. Must be willing and able to undergo bone marrow aspirates per protocol (with or without bone marrow biopsy per institutional guidelines). The bone marrow aspirate/biopsy must be adequate to allow for comparison for the on-study efficacy assessments.
9. Females of childbearing potential (FCBP) - An FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

1. Prior histone deacetylase (HDAC), dichloroacetate (DAC), or valproic acid for the treatment of cancer
2. Prior treatment with carfilzomib
3. Daily requirement for corticosteroids > prednisone 10 mg/day or equivalent
4. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the Principal Investigator prior to enrollment)
   * History of congenital long QT syndrome
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as heart rate (HR) < 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
   * ECG evidence of acute ischemia or grade 3 conduction system abnormalities (unless subject has a pacemaker)
   * Screening ECG with a corrected QT interval (QTc) > 450 msec
   * Right bundle branch block + left anterior hemiblock (bifascicular block)
   * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
   * Other clinically significant heart disease (e.g., congestive heart failure [CHF] New York Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen) (Patients with a history of atrial arrhythmias may be eligible if they are controlled and approved by the Lead Principal Investigator)
6. Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat. Inability to take oral medications, requirement for IV alimentation, active peptic ulcer disease or prior surgical procedures or bowel resection affecting absorption of oral medications.
7. Patients with diarrhea > Common Toxicity Criteria for Adverse Effects (CTCAE) grade 1 (increase of 4 stools per day over baseline mild increase in ostomy output compared to baseline)
8. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
9. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug [allow 72 hour washout period]
10. Concomitant use of cytochrome P450 3A4 (CYP3A4) inhibitors
11. Patients who have received either vaccine or antibody based therapy within ≤ 8 weeks; chemotherapy within ≤ 4 weeks, immunomodulatory drugs (IMiDs) within 2 weeks; or radiation therapy to > 30% of marrow-bearing bone within ≤ 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies
12. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
13. Peripheral blood stem cell transplant within 12 weeks of first dose of study treatment
14. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control
15. Male patients whose sexual partners are FCBP not using effective birth control
16. Patients with a prior malignancy with in the last 3 years (except for basal or squamous cell carcinoma, or in situ cancer or low risk prostate cancer after curative therapy or with > 90% remission at 5 years)
17. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
18. Significant neuropathy (≥ grade 3 or grade 2 with pain) within 14 days of initiation of therapy
19. Subjects with evidence of mucosal or internal bleeding, an active bleeding diathesis and or known platelet transfusion refractoriness
20. Patients with contraindications to any of the required concomitant drugs or supportive treatments, including hypersensitivity to anticoagulation and antiplatelet options, antiviral drugs, or tolerance to hydration due to pre-existing pulmonary of cardiac impairment
21. Patients with hypersensitivity to any of the components of the drug including allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib), including voriconazole, ziprasidone, aripiprazole and amiodarone
22. Ongoing graft-versus-host disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of the combination of panobinostat and carfilzomib | 28 day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kaufman, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Result] Kaufman JL, Mina R, Jakubowiak AJ, Zimmerman TL, Wolf JJ, Lewis C, Gleason C, Sharp C, Martin T, Heffner LT, Nooka AK, Harvey RD, Lonial S. Combining carfilzomib and panobinostat to treat relapsed/refractory multiple myeloma: results of a Multiple Myeloma Research Consortium Phase I Study. Blood Cancer J. 2019 Jan 4;9(1):3. doi: 10.1038/s41408-018-0154-8. PMID 30610196